CLINICAL TRIAL: NCT01200394
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP, MULTI-CENTER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF ONCE-DAILY ADMINISTRATION OF A PHOSPHODIESTERASE 5 INHIBITOR (PF-00489791) IN ADULTS WITH TYPE 2 DIABETES AND OVERT NEPHROPATHY
Brief Title: A Phase 2, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of PF-00489791 In Patients With Type 2 Diabetes And Overt Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7331011; 2010-021358-20 (EudraCT Number)
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetic nephropathy; chronic kidney disease; PF-00489791; phosphodiesterase; PDE5
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic | interventions — PF-00489791

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-00489791 (Experimental)
  Interventions: Drug: PF-00489791
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-00489791 — Tablet, 20 mg once daily for 12 weeks
  Arms: PF-00489791
Drug: Placebo — Tablet, placebo once daily for 12 weeks
  Arms: Placebo

SUMMARY:
PF-00489791 is an inhibitor of phosphodiesterase type 5. Our hypothesis is that PF-00489791 will enhance the relaxation of blood vessels within the kidney and so reduce blood pressure, improving renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects greater than or equal to 18 years. Female subjects must be of non-child bearing potential.
* Clinical diagnosis of type 2 diabetes together with stages 3a, 3b or 4 CKD, based on an eGFR of 25-59 mL/min/1.73m2.
* Evidence of persistent, overt albuminuria; defined as a UACR greater than or equal to 300 mg/g (greater than or equal to 33.9 mg/mmol) for greater than 3 months.

Exclusion Criteria:

* Subjects with CKD resulting from type 1 diabetes or non-diabetic CKD.
* Subjects with poorly controlled diabetes mellitus, defined as HbA1C >9%.
* Subjects on combination ACE inhibitor/ARB therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (159):
- United States (62):
  - Saadat Ansari Internal Medicine, Huntsville, Alabama
  - The Office of Iqbal Saeed MD, LLC, Huntsville, Alabama
  - AKDHC Medical Research Services, LLC*, Glendale, Arizona
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - North America Research Institute, Azusa, California
  - North American Research Institute / California Kidney Specialist, Azusa, California
  - Citrus Dialysis Center, Covina, California
  - California Institute of Renal Research, La Mesa, California
  - Capital Nephrology Clinical Research, Sacramento, California
  - California Kidney Specialists, San Dimas, California
  - American Institute of Research, Whittier, California
  - Whittier Internal Medicine Nephrology Medical Group, Whittier, California
  - North Valley Nephrology, Yuba City, California
  - Riverside Clinical Research, Edgewater, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - ASA Clinical Research, LLC, Jupiter, Florida
  - Lakeview Medical Research, Summerfield, Florida
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Renal Physicians of Georgia, Macon, Georgia
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Associates in Nephrology, SC, Evergreen Park, Illinois
  - Research by Design, LLC, Evergreen Park, Illinois
  - RenalCare Associates, Peoria, Illinois
  - Investigative Clinical Research of Indiana, LLC, Elwood, Indiana
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Biolab Research, LLC, Rockville, Maryland
  - Alzohaili Medical Consultants, Dearborn, Michigan
  - Apex Medical Research, AMR, Inc., Flint, Michigan
  - Apex Medical Research, MI, Inc., Flint, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Lincoln Nephrology and Hypertension, Lincoln, Nebraska
  - Nebraska Nephrology Research Institute, LLC - Research Management, Inc., Lincoln, Nebraska
  - Alliance Against Diabetes, Las Vegas, Nevada
  - Clinical Research Consortium, Las Vegas, Nevada
  - Jacobi Medical Center - Department of Medicine - Nephrology, The Bronx, New York
  - Mountain Kidney and Hypertension Associates, PA, Asheville, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Lake Medical Research, Willoughby Hills, Ohio
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Uniontown, Pennsylvania
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Carolina Nephrology, PA, Greenville, South Carolina
  - Palmetto Nephrology, PA, Orangeburg, South Carolina
  - South Carolina Nephrology & Hypertension Ctr, Inc, Orangeburg, South Carolina
  - South Carolina Nephrology and Hypertension Center, Orangeburg, South Carolina
  - Central Texas Kidney Associates, Austin, Texas
  - Research Management, Inc., Austin, Texas
  - Diagnostic Clinic of Houston, PA, Houston, Texas
  - Houston Nephrology Research, Houston, Texas
  - Research Across America, Houston, Texas
  - Renal Associates, PA, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, P.L.L.C., San Antonio, Texas
  - Nephrology Associates of Northern Virginia, Inc., Fairfax, Virginia
  - Nephrology Specialists, P.C., Mechanicsville, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Renal Remission & Hypertension Consultants, PLLC, Bremerton, Washington
  - Sound Medical Research, Port Orchard, Washington
  - Renal Remission and Hypertension Clinic, Silverdale, Washington
- Australia (5):
  - Renal Research Practice, Gosford, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Department of Nephrology, New Lambton, Newcastle
  - Pharmacy Department, New Lambton, Newcastle
  - Melbourne Renal Research Group, Reservoir, Victoria
- Canada (14):
  - Sheldon M Chumir Health Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Entralogix Clincal Research Inc., Brampton, Ontario
  - Entralogix Clinical Research Inc., Brampton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Entralogix Clinical Research Inc., Oakville, Ontario
  - N/A - formerly with Entralogix SMO, Toronto, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Centre de sante et de services sociaux champlain-Charles-Le Moyne, Greenfield Park, Quebec
  - Centre de Dialyse de Bois de Boulogne, Montreal, Quebec
  - Hopital de Sacre Coeur de Montreal, Montreal, Quebec
  - Saskatoon Nephrology Group, Nurses Redisence, Saskatoon, Saskatchewan
  - Saskatoon Nephrology Group, Nurses Residence, Saskatoon, Saskatchewan
  - Saskatoon Nephrology Group, Saskatoon, Saskatchewan
- Denmark (3):
  - Aarhus Universitetshospital (Aarhus Sygehus), Aarhus
  - Rigshospitalet, Copenhagen Oe
  - Steno Diabetes Center, Gentofte Municipality
- Hong Kong (5):
  - Queen Mary Hospital, Hong Kong
  - Division of Nephrology, Dept. of Medicine, Pokfulam
  - Division of Nephrology, Pokfulam
  - ICON Clinical Research, Quarry Bay
  - Prince of Wales Hospital, Shatin
- India (10):
  - Apollo Hospitals, Hyderabad, Andhra Pradesh
  - Gujarat Kidney Foundation, Ahmedabad, Gujarat
  - Shrushrut Clinical Research Association, Ahmedabad, Gujarat
  - P. D. Hinduja National Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Pfizer Centre, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Diabetes Care and Research Centre, Pune, Maharashtra
  - KE.M Hospital Research Centre, Pune, Maharashtra
  - King Edward Memorial Hospital, Pune, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
- Malaysia (7):
  - Universiti Sains Malaysia, Kota Bharu, Kelantan
  - Unit Kajian Klinikal, Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Taiping, Taiping, Perak
  - Clinical Research Centre, Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Nephrology Clinic, Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Unit Hemodialisis, Hospital Serdang, Kajang, Selangor
- Mexico (5):
  - ICLE SC, Guadalajara, Jalisco
  - Comite Mexicano para la Prevencion de la Osteoporosis, A.C., Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (INCMNSZ), Tlalpan, Mexico City
  - Hospital Central Dr Ignacio Morones Prieto Unidad Regional de Osteoporosis, San Luis Potosí City, San Luis Potosí
  - Hospital Angeles del Pedregal, Angeles Del Pedregal Cp.
- Poland (9):
  - NZOZ "DIAGNOMED" S.C., Poradnia Nefrologiczna, Bielsko-Biala
  - Samodzielny Publiczny Szpital Kliniczny im Andrzeja Mieleckiego, Katowice
  - NZOZ PS "Medica", Lublin
  - Centrum Medyczne "Osteomed" NZOZ, Lecznica Specjalistow, Warsaw
  - Centrum Medyczne "OSTEOMED" NZOZ, Warsaw
  - Centrum Medyczne "Osteomed", Warsaw
  - Centrum Medyczne OSTEOMED NZOZ; Lecznica Specjalistaw, Warsaw
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - SPZOZ Akademicki Szpital Kliniczny im. J. Mikulicza - Radeckiego, Wroclaw
- Serbia (6):
  - Clinical Center of Serbia Institute for Endocrinology, Diabetes and Metabolic Diseases, Belgrade
  - Clinic for Nephrology, Military Medical Academy, Belgrade
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center "Zvezdara", Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Clinic for Endocrinology, Clinical Center Nis, Niš
- Slovakia (4):
  - FNsP Bratislava, Nemocnica Stare Mesto, Bratislava
  - Nemocnice s poliklinikami n.o., Levice
  - Fakultna nemocnica s poliklinikou J.A.Reimana Presov, Prešov
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
- South Africa (11):
  - Worthwhile Clinical Trials (WWCT), Lake View Hospital, Benoni, Gauteng
  - Dr. George Mukhari Hospital -University of Limpopo, Pretoria, Gauteng
  - Wits Clinical research, Johannesburg, Gauteng- South Africa
  - Centre for Diabetes and Endocrinology, Durban, KwaZulu-Natal
  - Latros International, Bloemfontein
  - Division of Nephrology and Hypertension, E13 Renal Unit, Cape Town
  - St Augustine's Hospital, Durban
  - Centre for Diabetes and Endocrinology, Durban
  - Centre for Diabetes and Endocrinology, Houghton, Johannesburg
  - Intercare Parow Medical and Dental Centre, Parow
  - Medi-Clinic Heart Hospital (Pretoria Heart Hospital), Pretoria
- South Korea (9):
  - Pharmacy, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Clinical Trial Pharmacy, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Department of Pharmacy, Seoul
  - Samsung Medical Center,Sungkyunkwan Univ School of Medicine, Seoul
  - Samsung Medical Center/Division of Nephrology, Seoul
  - Boramae Medical Center/Division of Nephrology, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Sweden (3):
  - Sahlgrenska University Hospital Njurmottagningen, Gothenburg
  - A+ Science City site, Stockholm
  - Akademiska Sjukhuset, Uppsala
- United Kingdom (6):
  - Doncaster Royal Infirmary, Doncaster, South Yorkshire
  - Research Offices (5th Floor), Coventry
  - University of Edinburgh, Edinburgh
  - The Royal London Hospital Whitechapel, London
  - Guy's and St Thomas' Foundation Trust, London
  - Northern General Hospital Campus, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7331011&StudyName=A%20Phase%202%2C%20Placebo-Controlled%20Study%20To%20Evaluate%20The%20Efficacy%20And%20Safety%20Of%20PF-00489791%20In%20Patients%20With%20Type%202%20Diabetes%20And%20Overt%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to PF-00489791 tablet orally once daily for 12 weeks.
- PF-00489791 20 mg: PF-00489791 20 milligram (mg) tablet orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-00489791 20 mg
Started | 64 | 192
Completed | 62 | 164
Not Completed | 2 | 28
Not completed — Adverse Event | 0 | 14
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did Not Meet Entrance Criteria | 1 | 4
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication and had at least 1 post-dose efficacy measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-00489791 20 mg | Total
Number analyzed (Participants) | 64 | 192 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.0) | 62.0 (8.8) | 61.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 48 | 61
  Male | 51 | 144 | 195
Race/Ethnicity, Customized [Number; unit: participants]
  White | 27 | 79 | 106
  Black | 5 | 13 | 18
  Asian | 26 | 83 | 109
  Other | 6 | 17 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urinary Albumin Creatinine Ratio (UACR) at Week 12
Description: UACR was ratio of albumin measured in urine (milligram) to creatinine measured in urine (millimole), reported in units milligram per millimole (mg/mmol). A decrease in UACR may be associated with improved renal and cardiovascular function. The mean values of the 3 consecutive first morning void urine samples (obtained 2 days prior to [Day 5, 6 of Week 12], and with last sample collected on the morning of scheduled clinic visit [Day 7 of Week 12]) were used to determine UACR at the scheduled clinic visit. The mean values of the 3 consecutive first morning void urine samples obtained at screening were used to determine baseline UACR.
Time Frame: Baseline, Week 12 (Day 5, 6, 7)
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication and had at least 1 post-dose efficacy measurement. Here, 'Number analyzed' = Participants evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
mg/mmol
  Baseline: number analyzed (Participants) | 63 | 191
  Baseline | 195.130 (171.8116) | 182.378 (156.5097)
  Change at Week 12: number analyzed (Participants) | 60 | 164
  Change at Week 12 | 9.072 (176.4360) | -6.539 (128.4866)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 20 mg; Analysis of covariance (ANCOVA) model within an outlier robust Bayesian framework on normal logarithmic scale with treatment as fixed effect, baseline UACR and baseline supine systolic blood pressure (BP) as covariate. Values were back-transformed from log scale. Model used informative prior distribution for placebo; Test type: Superiority; p = 0.9889, ANCOVA — Posterior distribution was used to calculate a probability (presented as P-value) that PF-00489791 has a greater than 0% reduction in UACR compared to placebo; Geometric Mean Ratio = 0.843, 95% CI 2-sided [0.728 to 0.975] — Geometric mean ratio and corresponding 95% credible intervals were calculated
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 20 mg; ANCOVA model within an outlier robust Bayesian framework on normal logarithmic scale with treatment as fixed effect, baseline UACR and baseline supine systolic BP as covariate. Values were back-transformed from log scale. Model used informative prior distribution for placebo; Test type: Superiority; p = 0.2402, ANCOVA — Posterior distribution was used to calculate a probability (presented as P-value) that PF-00489791 has a greater than or equal to 20% reduction in UACR compared to placebo

2. Secondary Outcome: Change From Baseline in Urinary Albumin Creatinine Ratio (UACR) at Week 3, 6 and 16
Description: UACR was ratio of albumin measured in urine (milligram) to creatinine measured in urine (millimole), reported in units mg/mmol. A decrease in UACR may be associated with improved renal and cardiovascular function. The mean values of the 3 consecutive first morning void urine samples (obtained 2 days prior to [Day 5, 6 of specified Week], and with last sample collected on the morning of scheduled clinic visit [Day 7 of specified Week]) were used to determine UACR at the scheduled clinic visit. The mean values of the 3 consecutive first morning void urine samples obtained at screening were used to determine baseline UACR.
Time Frame: Baseline, Week 3 (Day 5, 6, 7), Week 6 (Day 5, 6, 7), Week 16 (Day 5, 6, 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
mg/mmol
  Change at Week 3: number analyzed (Participants) | 60 | 171
  Change at Week 3 | -11.805 (161.7282) | -14.268 (94.8469)
  Change at Week 6: number analyzed (Participants) | 62 | 171
  Change at Week 6 | -7.772 (162.0838) | -2.546 (179.5896)
  Change at Week 16: number analyzed (Participants) | 60 | 162
  Change at Week 16 | 16.500 (202.7600) | 2.802 (107.9582)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 20 mg; Week 3: Mixed model repeated measures (MMRM) on normal logarithmic scale with baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.0382, Mixed Models Analysis; Geometric Mean Ratio = 0.8759, 95% CI 2-sided [0.7727 to 0.9927]
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 20 mg; Week 6: MMRM on normal logarithmic scale with baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.0112, Mixed Models Analysis; Geometric Mean Ratio = 0.8311, 95% CI 2-sided [0.7208 to 0.9584]
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20 mg; Week 16: MMRM on normal logarithmic scale with baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.1490, Mixed Models Analysis; Geometric Mean Ratio = 0.8816, 95% CI 2-sided [0.7427 to 1.0465]

3. Secondary Outcome: Change From Baseline in Urinary Protein Creatinine Ratio (UPCR) at Week 3, 6, 12, and 16
Description: UPCR is a ratio between two measured substances in urine: milligram of protein per millimole (mmol) of creatinine, reported in units mg/mmol. A decrease in UPCR may be associated with improved renal and cardiovascular function. The mean values of the 3 consecutive first morning void urine samples (obtained 2 days prior to [Day 5, 6 of Week 3, 6, 12, 16], and with last sample collected on the morning of scheduled clinic visit [Day 7 of Week 3, 6, 12, 16]) were used to determine UPCR at the scheduled clinic visit. The mean values of the 3 consecutive first morning void urine samples obtained at screening were used to determine baseline UPCR.
Time Frame: Baseline, Week 3 (Day 5, 6, 7), Week 6 (Day 5, 6, 7), Week 12 (Day 5, 6, 7), Week 16 (Day 5, 6, 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
mg/mmol
  Baseline: number analyzed (Participants) | 63 | 191
  Baseline | 282.208 (259.8496) | 261.015 (220.5260)
  Change at Week 3: number analyzed (Participants) | 60 | 170
  Change at Week 3 | -20.302 (247.4490) | -26.883 (161.0038)
  Change at Week 6: number analyzed (Participants) | 62 | 170
  Change at Week 6 | -10.278 (256.7216) | 10.699 (290.5749)
  Change at Week 12: number analyzed (Participants) | 59 | 164
  Change at Week 12 | 14.632 (283.9874) | -5.371 (207.3333)
  Change at Week 16: number analyzed (Participants) | 60 | 162
  Change at Week 16 | 30.880 (332.0766) | 20.299 (190.3546)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 20 mg; Week 3: MMRM on normal logarithmic scale with baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.0297, Mixed Models Analysis; Geometric Mean Ratio = 0.8565, 95% CI 2-sided [0.7450 to 0.9847]
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 20 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0305, Mixed Models Analysis; Geometric Mean Ratio = 0.8524, 95% CI 2-sided [0.7376 to 0.9850]
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20 mg; Week 12: MMRM on normal logarithmic scale with baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.0068, Mixed Models Analysis; Geometric Mean Ratio = 0.7937, 95% CI 2-sided [0.6717 to 0.9378]
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 20 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.1151, Mixed Models Analysis; Geometric Mean Ratio = 0.8634, 95% CI 2-sided [0.7190 to 1.0368]

4. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 3, 6, 12, and 16
Description: The eGFR was calculated using 4 variable formula developed by the modification of diet in renal disease (MDRD) study group. The 4 variables needed to estimate glomerular filtration rate (GFR) using this formula were serum creatinine concentration (sCr), age, sex (for females, eGFR was multiplied by 0.742) and ethnic origin (for African-Caribbean people only, eGFR was multiplied by 1.212). Thus eGFR in milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) = 175*(sCr/88.4)^-1.154*(Age)^-0.203*(0.742 if female)*(1.212 if African-Caribbean). Baseline eGFR was determined predose at Week 0 (Day 1).
Time Frame: Baseline, Week 3, 6, 12, 16 (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
mL/min/1.73 m^2
  Baseline: number analyzed (Participants) | 61 | 188
  Baseline | 38.575 (11.9122) | 37.740 (9.8834)
  Change at Week 3: number analyzed (Participants) | 59 | 172
  Change at Week 3 | 0.069 (6.2868) | -0.156 (4.6044)
  Change at Week 6: number analyzed (Participants) | 59 | 166
  Change at Week 6 | -0.930 (5.3513) | -0.755 (5.2701)
  Change at Week 12: number analyzed (Participants) | 58 | 161
  Change at Week 12 | -1.435 (5.3757) | -1.463 (5.1074)
  Change at Week 16: number analyzed (Participants) | 59 | 163
  Change at Week 16 | -1.915 (5.9005) | -1.659 (6.0659)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 20 mg; Week 3: MMRM on normal logarithmic scale with change from baseline as response variable and baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.3585, Mixed Models Analysis; Geometric Mean Ratio = 0.9816, 95% CI 2-sided [0.9434 to 1.0214]
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 20 mg; Week 6: MMRM on normal logarithmic scale with change from baseline as response variable and baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.7475, Mixed Models Analysis; Geometric Mean Ratio = 0.9939, 95% CI 2-sided [0.9577 to 1.0315]
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20 mg; Week 12: MMRM on normal logarithmic scale with change from baseline as response variable and baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.4972, Mixed Models Analysis; Geometric Mean Ratio = 0.9866, 95% CI 2-sided [0.9488 to 1.0259]
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 20 mg; Week 16: MMRM on normal logarithmic scale with change from baseline as response variable and baseline, baseline supine systolic BP, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. Unstructured covariance matrix was used to estimate variances and covariance within participant across time points. Values were back-transformed from log scale; Test type: Superiority; p = 0.9146, Mixed Models Analysis; Geometric Mean Ratio = 1.0024, 95% CI 2-sided [0.9588 to 1.0481]

5. Secondary Outcome: Systolic, Diastolic and Mean Blood Pressure at Week 0, 3, 6, 12, and 16
Description: Systolic blood pressure (SBP) is the blood pressure (pressure exerted by circulating blood on the walls of blood vessels) when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle of heart. diastolic blood pressure (DBP) is the blood pressure (pressure exerted by circulating blood on the walls of blood vessels) when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles of heart. Mean blood pressure (MBP) = diastolic blood pressure + ([systolic blood pressure - diastolic blood pressure]/3). After a minimum of 5 minutes of rest, supine BP was measured with the participant's arm supported at the level of the heart.
Time Frame: Week 0, 3, 6, 12, 16 (follow-up)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
millimeter of mercury (mmHg)
  Supine Systolic BP, Week 0 | 137.20 [135.01 to 139.40] | 131.81 [130.53 to 133.10]
  Supine Diastolic BP, Week 0 | 76.98 [75.53 to 78.42] | 73.27 [72.43 to 74.11]
  Supine Mean BP, Week 0 | 107.27 [105.66 to 108.88] | 102.68 [101.74 to 103.62]
  Supine Systolic BP, Week 3 | 136.68 [134.30 to 139.05] | 136.15 [134.74 to 137.56]
  Supine Diastolic BP, Week 3 | 76.78 [75.25 to 78.31] | 77.18 [76.27 to 78.10]
  Supine Mean BP, Week 3 | 107.06 [105.32 to 108.80] | 106.90 [105.86 to 107.94]
  Supine Systolic BP, Week 6 | 137.41 [134.90 to 139.93] | 136.94 [135.42 to 138.45]
  Supine Diastolic BP, Week 6 | 76.88 [75.32 to 78.43] | 76.41 [75.48 to 77.35]
  Supine Mean BP, Week 6 | 107.37 [105.58 to 109.15] | 106.70 [105.62 to 107.77]
  Supine Systolic BP, Week 12 | 136.89 [133.73 to 140.06] | 137.70 [135.79 to 139.60]
  Supine Diastolic BP, Week 12 | 77.32 [75.51 to 79.13] | 76.69 [75.61 to 77.78]
  Supine Mean BP, Week 12 | 107.41 [105.27 to 109.55] | 107.14 [105.85 to 108.42]
  Supine Systolic BP, Week 16 | 138.38 [135.51 to 141.25] | 138.89 [137.15 to 140.63]
  Supine Diastolic BP, Week 16 | 77.25 [75.59 to 78.92] | 77.90 [76.90 to 78.91]
  Supine Mean BP, Week 16 | 108.00 [106.10 to 109.91] | 108.47 [107.31 to 109.62]
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 20 mg; Supine Systolic BP, Week 0: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares (LS) Mean Difference = -5.39, 95% CI 2-sided [-7.94 to -2.84], Standard Error of Mean 1.2942
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 20 mg; Supine Diastolic BP, Week 0: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -3.71, 95% CI 2-sided [-5.38 to -2.04], Standard Error of Mean 0.8490
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20 mg; Supine Mean BP, Week 0: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -4.59, 95% CI 2-sided [-6.46 to -2.72], Standard Error of Mean 0.9489
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 20 mg; Supine Systolic BP, Week 3: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.7093, Mixed Models Analysis; LS Mean Difference = -0.52, 95% CI 2-sided [-3.29 to 2.24], Standard Error of Mean 1.4056
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; Supine Diastolic BP, Week 3: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.6564, Mixed Models Analysis; LS Mean Difference = 0.40, 95% CI 2-sided [-1.39 to 2.20], Standard Error of Mean 0.9089
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 20 mg; Supine Mean BP, Week 3: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.8763, Mixed Models Analysis; LS Mean Difference = -0.16, 95% CI 2-sided [-2.20 to 1.87], Standard Error of Mean 1.0334
Statistical Analysis 7: Comparison: Placebo vs PF-00489791 20 mg; Supine Systolic BP, Week 6: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.7491, Mixed Models Analysis; LS Mean Difference = -0.48, 95% CI 2-sided [-3.42 to 2.46], Standard Error of Mean 1.4926
Statistical Analysis 8: Comparison: Placebo vs PF-00489791 20 mg; Supine Diastolic BP, Week 6: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.6141, Mixed Models Analysis; LS Mean Difference = -0.47, 95% CI 2-sided [-2.29 to 1.35], Standard Error of Mean 0.9235
Statistical Analysis 9: Comparison: Placebo vs PF-00489791 20 mg; Supine Mean BP, Week 6: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.5281, Mixed Models Analysis; LS Mean Difference = -0.67, 95% CI 2-sided [-2.75 to 1.42], Standard Error of Mean 1.0582
Statistical Analysis 10: Comparison: Placebo vs PF-00489791 20 mg; Supine Systolic BP, Week 12: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.6695, Mixed Models Analysis; LS Mean Difference = 0.80, 95% CI 2-sided [-2.90 to 4.50], Standard Error of Mean 1.8764
Statistical Analysis 11: Comparison: Placebo vs PF-00489791 20 mg; Supine Diastolic BP, Week 12: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.5607, Mixed Models Analysis; LS Mean Difference = -0.63, 95% CI 2-sided [-2.74 to 1.49], Standard Error of Mean 1.0730
Statistical Analysis 12: Comparison: Placebo vs PF-00489791 20 mg; Supine Mean BP, Week 12: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.8297, Mixed Models Analysis; LS Mean Difference = -0.27, 95% CI 2-sided [-2.78 to 2.23], Standard Error of Mean 1.2722
Statistical Analysis 13: Comparison: Placebo vs PF-00489791 20 mg; Supine Systolic BP, Week 16: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.7644, Mixed Models Analysis; LS Mean Difference = 0.51, 95% CI 2-sided [-2.85 to 3.87], Standard Error of Mean 1.7065
Statistical Analysis 14: Comparison: Placebo vs PF-00489791 20 mg; Supine Diastolic BP, Week 16: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.5123, Mixed Models Analysis; LS Mean Difference = 0.65, 95% CI 2-sided [-1.30 to 2.61], Standard Error of Mean 0.9917
Statistical Analysis 15: Comparison: Placebo vs PF-00489791 20 mg; Supine Mean BP, Week 16: MMRM model included baseline, visit, treatment, baseline by visit interaction and treatment by visit interaction as fixed effects. The unstructured covariance matrix was used to estimate variances and covariance within participant across time points; Test type: Superiority; p = 0.6838, Mixed Models Analysis; LS Mean Difference = 0.46, 95% CI 2-sided [-1.77 to 2.70], Standard Error of Mean 1.1355

6. Secondary Outcome: Change From Baseline in Serum Creatinine Concentration at Week 3, 6, 12, and 16
Description: Serum creatinine concentration was used as a marker of renal function. Baseline serum creatinine concentration was determined predose at Week 0 (Day 1).
Time Frame: Baseline, Week 3, 6, 12, 16 (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
micromole per liter (mcmol/L)
  Baseline: number analyzed (Participants) | 61 | 188
  Baseline | 164.929 (42.0837) | 163.637 (42.9529)
  Change at Week 3: number analyzed (Participants) | 59 | 172
  Change at Week 3 | 1.232 (23.9961) | 2.691 (20.6884)
  Change at Week 6: number analyzed (Participants) | 59 | 166
  Change at Week 6 | 3.158 (18.0835) | 4.974 (21.7977)
  Change at Week 12: number analyzed (Participants) | 58 | 161
  Change at Week 12 | 6.139 (20.7198) | 8.110 (22.3709)
  Change at Week 16: number analyzed (Participants) | 59 | 163
  Change at Week 16 | 11.527 (28.5175) | 9.269 (26.6470)

7. Secondary Outcome: Change From Baseline in Urine Transforming Growth Factor (TGF) Beta-1 Concentration at Week 3, 6, 12, and 16
Description: TGF Beta-1 is a major fibrogenic growth factor implicated in the pathogenesis of renal scarring. It is overexpressed in the diabetic kidney where it may promote matrix accumulation. Baseline TGF Beta-1 concentration was determined predose at Week 0 (Day 1).
Time Frame: Baseline, Week 3, 6, 12, 16 (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
picogram per milliliter (pg/mL)
  Baseline: number analyzed (Participants) | 55 | 159
  Baseline | 177.88 (231.154) | 213.37 (274.409)
  Change at Week 3: number analyzed (Participants) | 52 | 145
  Change at Week 3 | -22.81 (260.140) | -54.06 (349.817)
  Change at Week 6: number analyzed (Participants) | 53 | 141
  Change at Week 6 | 23.33 (345.304) | -68.59 (333.378)
  Change at Week 12: number analyzed (Participants) | 49 | 136
  Change at Week 12 | -36.20 (281.523) | -11.87 (328.482)
  Change at Week 16: number analyzed (Participants) | 49 | 125
  Change at Week 16 | -23.54 (134.752) | -31.32 (299.546)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.5422, Mixed Models Analysis; Geometric Mean Ratio = 0.9282, 95% CI 2-sided [0.7297 to 1.1807]
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 20 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0490, Mixed Models Analysis; Geometric Mean Ratio = 0.7998, 95% CI 2-sided [0.6402 to 0.9990]
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.7264, Mixed Models Analysis; Geometric Mean Ratio = 1.0435, 95% CI 2-sided [0.8211 to 1.3262]
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 20 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 0.3733, Mixed Models Analysis; Geometric Mean Ratio = 1.1154, 95% CI 2-sided [0.8761 to 1.4201]

8. Secondary Outcome: Change From Baseline in Serum High Sensitivity C-Reactive Protein (Hs-CRP) Concentration at Week 12 and 16
Description: The CRP is an acute phase reactant which is virtually absent from the blood serum of healthy persons but rapidly appears in blood and body fluids in response to injurious stimuli. Baseline hs-CRP was determined predose at Week 0 (Day 1).
Time Frame: Baseline, Week 12, 16 (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
milligram per liter (mg/L)
  Baseline: number analyzed (Participants) | 60 | 187
  Baseline | 3.019 (3.4924) | 4.330 (8.6809)
  Change at Week 12: number analyzed (Participants) | 56 | 160
  Change at Week 12 | 1.183 (3.4600) | 0.106 (7.4909)
  Change at Week 16: number analyzed (Participants) | 57 | 161
  Change at Week 16 | 0.317 (2.9508) | -0.102 (6.3317)

9. Secondary Outcome: Change From Baseline in Serum Cystatin-C Concentration at Week 12 and 16
Description: Cystatin C is produced by all nucleated cells at a constant rate and is freely filtered at the glomerulus. The blood concentration of cystatin C depends almost entirely on the GFR and is not substantially affected by diet, nutritional status or inflammatory disease. Serum cystatin C had been proposed as an endogenous marker of GFR in participant with chronic kidney disease (CKD) than sCr. Baseline serum cystatin C was determined predose at Week 0 (Day 1).
Time Frame: Baseline, Week 12, 16 (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
mg/L
  Baseline: number analyzed (Participants) | 60 | 188
  Baseline | 1.659 (0.4122) | 1.695 (0.4497)
  Change at Week 12: number analyzed (Participants) | 56 | 161
  Change at Week 12 | 0.096 (0.1844) | 0.070 (0.2890)
  Change at Week 16: number analyzed (Participants) | 57 | 162
  Change at Week 16 | 0.104 (0.3234) | 0.075 (0.3176)

10. Secondary Outcome: Plasma Concentration Versus Time Summary of PF-00489791
Time Frame: Pre-dose at Day 1 of Week 0, 3, 6 and 12; 4 hours post-dose on Day 1 of Week 0, 3 and 6
Population: Pharmacokinetic analysis set included all randomized and treated participants with at least 1 measured PF-00489791 concentration. Here, "Number analyzed" signifies number of participants evaluable for specified categories. This outcome measure was planned not to be analyzed for Placebo reporting arm.
Measure: Mean (Standard Deviation); unit: microgram per millilitre (microgram/mL)
Arm/Group | PF-00489791 20 mg
Number analyzed (Participants) | 191
microgram per millilitre (microgram/mL)
  4 hours post-dose at Day 1 of Week 0: number analyzed (Participants) | 189
  4 hours post-dose at Day 1 of Week 0 | 0.6540 (0.33644)
  Pre-dose at Day 1 of Week 3: number analyzed (Participants) | 164
  Pre-dose at Day 1 of Week 3 | 0.4156 (0.44674)
  4 hours post-dose at Day 1 of Week 3: number analyzed (Participants) | 166
  4 hours post-dose at Day 1 of Week 3 | 0.9772 (0.59610)
  Pre-dose at Day 1 of Week 6: number analyzed (Participants) | 164
  Pre-dose at Day 1 of Week 6 | 0.3514 (0.40417)
  4 hours post-dose at Day 1 of Week 6: number analyzed (Participants) | 165
  4 hours post-dose at Day 1 of Week 6 | 0.9274 (0.52405)
  Pre-dose at Day 1 of Week 12: number analyzed (Participants) | 162
  Pre-dose at Day 1 of Week 12 | 0.3930 (0.41593)

11. Other Pre Specified Outcome: Change From Baseline in Plasma Glycosylated Hemoglobin (HbA1c) Level at Week 12 and 16
Description: Level of HbA1c is an indicator for the average level of blood glucose over the previous 3 months. Baseline HbA1c level was determined predose at Week 0 (Day 1).
Time Frame: Baseline, Week 12, 16 (follow-up)
Population: Safety analysis set consists of all participants who received at least 1 dose of study medication. Here, 'Number analyzed' = Participants evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
percentage of hemoglobin
  Baseline: number analyzed (Participants) | 61 | 187
  Baseline | 7.13 (1.023) | 7.39 (1.135)
  Change at Week 12: number analyzed (Participants) | 56 | 157
  Change at Week 12 | 0.12 (0.856) | -0.28 (0.975)
  Change at Week 16: number analyzed (Participants) | 58 | 161
  Change at Week 16 | 0.14 (1.009) | -0.09 (0.986)

12. Other Pre Specified Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for determining vital signs abnormalities: supine or standing systolic BP (SBP) (less than [<] 90 mmHg and increase or decrease of greater than or equal to [>=] 30 mmHg compared to baseline value), supine or standing diastolic BP (DBP) (<50 mmHg and increase or decrease of >=20 mmHg compared to baseline value), supine pulse rate (>120 beats per minute [bpm] or <40 bpm), standing pulse rate (>140 bpm or <40 bpm). For supine, baseline was the average of the triplicate predose readings at Week 0 (Day 1). For standing, baseline is the predose reading at Week 0 (Day 1). Only categories who had at least 1 participant are reported.
Time Frame: Baseline up to Week 16 (follow-up)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
Participants
  Supine SBP <90 mmHg | 0 | 1
  Standing SBP <90 mmHg: number analyzed (Participants) | 64 | 189
  Standing SBP <90 mmHg | 0 | 2
  Supine DBP <50 mmHg | 0 | 3
  Standing DBP <50 mmHg: number analyzed (Participants) | 64 | 189
  Standing DBP <50 mmHg | 0 | 3
  Supine Pulse Rate <40 bpm | 0 | 1
  Increase in Supine SBP >=30 mmHg | 0 | 14
  Increase in Standing SBP >=30 mmHg: number analyzed (Participants) | 64 | 189
  Increase in Standing SBP >=30 mmHg | 1 | 1
  Increase in Supine DBP >=20 mmHg | 0 | 7
  Increase in Standing DBP >=20 mmHg: number analyzed (Participants) | 64 | 189
  Increase in Standing DBP >=20 mmHg | 1 | 0
  Decrease in Supine SBP >=30 mmHg | 0 | 9
  Decrease in Standing SBP >=30 mmHg: number analyzed (Participants) | 64 | 189
  Decrease in Standing SBP >=30 mmHg | 2 | 11
  Decrease in Supine DBP >=20 mmHg | 0 | 5
  Decrease in Standing DBP >=20 mmHg: number analyzed (Participants) | 64 | 189
  Decrease in Standing DBP >=20 mmHg | 1 | 11

13. Other Pre Specified Outcome: Number of Participants With Edema and Fluid Overload
Description: Participants were assessed for signs of edema and fluid overload.
Time Frame: Week 0, 3, 6, 12, 16 (follow-up)
Population: Safety analysis set consists of all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
Participants
  Week 0 | 0 | 4
  Week 3 | 1 | 8
  Week 6 | 1 | 11
  Week 12 | 4 | 9
  Week 16 | 5 | 6

14. Other Pre Specified Outcome: Number of Participants With Increased Use of Diuretics
Time Frame: Baseline up to Week 16 (follow-up)
Population: Safety analysis set consists of all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
Participants | 3 | 10

15. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory test abnormalities: Hematology (hemoglobin [<0.8*lower limit of normal{LLN}], hematocrit [<0.8*LLN], red blood cells [<0.8*LLN], platelet [<0.5*LLN/>1.75*upper limit of normal{ULN}], white blood cells [<0.6*LLN/>1.5*ULN], lymphocytes [<0.8*LLN/>1.2*ULN], neutrophils [<0.8*LLN/>1.2*ULN], basophils [>1.2*ULN], eosinophils [>1.2*ULN], monocytes [>1.2*ULN]); Liver Function (total/direct/indirect bilirubin [>1.5*ULN], aspartate aminotransferase/ alanine aminotransferase/ gamma glutamyl transpeptidase/ lactate dehydrogenase/ alkaline phosphatase [>3.0*ULN]); Renal Function (blood urea nitrogen/ creatinine [>1.3*ULN], uric acid [>1.2*ULN]); Electrolytes (sodium [<0.95*LLN/>1.05*ULN], potassium, chloride, calcium, bicarbonate [<0.9*LLN/>1.1*ULN]); Clinical Chemistry (glucose [<0.6*LLN/>1.5*ULN], glycosylated hemoglobin [>1.3*ULN], Creatine Kinase [>2.0*ULN], Amylase, Lipase[>1.5*ULN]).
Time Frame: Baseline up to Week 16 (follow-up)
Population: Safety analysis set consists of all participants who received at least 1 dose of study medication. Here 'N' (Overall Number of Participants Analyzed) signifies participants evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 63 | 190
Participants | 62 | 190

16. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication and up to Week 16 (follow-up) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both non-serious (AEs) and serious adverse events (SAEs)
Time Frame: Baseline up to Week 16 (follow-up)
Population: Safety analysis set consists of all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 20 mg
Number analyzed (Participants) | 64 | 192
Participants
  AEs | 36 | 105
  SAEs | 6 | 13

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16 (follow-up)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. AEs included both non-serious (AEs) and serious adverse events (SAEs)
Arm/Group | Placebo | PF-00489791 20 mg
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/192
Serious Adverse Events (participants affected / at risk) | 6/64 | 13/192
Other Adverse Events (participants affected / at risk) | 35/64 | 104/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | PF-00489791 20 mg (N=192)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Prostatectomy (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | PF-00489791 20 mg (N=192)
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 2
Lacrimation increased (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 17
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 12
Flatulence (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 7
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Feeling hot (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 6 | 10
Pyrexia (General disorders) | 0 | 4
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1
Eye infection bacterial (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 3
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mastitis fungal (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 9
Onychomycosis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 6
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Amylase increased (Investigations) | 1 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 6
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose abnormal (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 3
Blood pressure abnormal (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 2
Blood uric acid increased (Investigations) | 2 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 2
Liver function test normal (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 7
Drooling (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 12
Memory impairment (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2
Polyuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Immobile (Social circumstances) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 9
Hypotension (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.